CLINICAL TRIAL: NCT03435627
Title: Post Marketing Surveillance on Long-term Use With Norditropin® (Short Stature Due to Noonan Syndrome)
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GHLIQUID-4358; U1111-1191-3084 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-01-31; First posted 2018-02-19 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Genetic Disorder; Noonan Syndrome
MeSH Terms: conditions — Genetic Diseases, Inborn; Noonan Syndrome | interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Norditropin® (naïve participants): The treatment period of Norditropin® for naïve participants will be up to 208 weeks.
  Interventions: Drug: Somatropin
- Norditropin® (non-naïve participants): The treatment period of Norditropin® for non-naïve participants will be up to 442 weeks.
  Interventions: Drug: Somatropin

INTERVENTIONS:
Drug: Somatropin — Participants will be treated with commercially available Norditropin® (somatropin) according to routine clinical practice at the discretion of the treating physician.

SUMMARY:
The purpose of this study is to collect information about safety and effectiveness for long term use of Norditropin®. Participants will attend the medical institution according to usual practice and receive medical care, as agreed with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
* The decision to initiate treatment with commercially available Norditropin® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study.
* For non-naïve patients; patients who were previously enrolled in study: GHLIQUID-4020.
* For naïve patients; short stature due to Noonan syndrome diagnosed by the physician and a decision to initiate treatment with Norditropin® has been made by the patient/parent and the physician. At study sites, all patients will be registered consecutively from the first patient after approval date (consecutively registered system).
* Male or female, 3 years old or over, bone age: less than 17 years old for male / less than 15 years old for female.

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Known or suspected allergy to study products or related products.
* In case of naïve patients, patients who have received growth hormone (GH) products for treatment of indication other than short stature due to Noonan syndrome before approval date of Noonan indication.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 60 patients (consisting of non-naïve patients who were previously enrolled in study: GHLIQUID-4020 and naïve patients enrolled after approval of the Noonan indication in Japan) are planned to be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Number of adverse drug reactions (ADR) | Weeks 0-208
  Count of events

SECONDARY OUTCOMES:
Number of serious adverse drug reaction (SADR) | Week 0-208
  Count of events
Number of serious adverse event (SAE) | Week 0-208
  Count of events
Number of cardiac adverse event (AE) | Week 0-208
  Count of events
Change in insulin like growth factor I (IGF-I) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Measured in ng/mL
Change in insulin like growth factor I (IGF-I) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Measured in ng/mL
Change in insulin like growth factor I standard deviation score (IGF-I SDS) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Presented as standard deviation (SD) score
Change in insulin like growth factor I standard deviation score (IGF-I SDS) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Presented as SD score
Change in haemoglobin A1c (HbA1c) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Measured in %
Change in haemoglobin A1c (HbA1c) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Measured in %
Change in aspartate aminotransferase (AST) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Measured in IU/L
Change in aspartate aminotransferase (AST) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Measured in IU/L
Change in alanine aminotransferase (ALT) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Measured in IU/L
Change in alanine aminotransferase (ALT) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Measured in IU/L
Change in total cholesterol (T-CHO) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Measured in mg/dL
Change in total cholesterol (T-CHO) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Measured in mg/dL
Change in high-density lipoprotein cholesterol (HDL-C) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Measured in mg/dL
Change in high-density lipoprotein cholesterol (HDL-C) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Measured in mg/dL
Change in Low-density lipoprotein cholesterol (LDL-C) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Measured in mg/dL
Change in Low-density lipoprotein cholesterol (LDL-C) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Measured in mg/dL
Change in triglyceride (TG) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Measured in mg/dL
Change in triglyceride (TG) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Measured in mg/dL
Change in thyroid stimulation hormone(TSH) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Measured in μU/mL
Change in thyroid stimulation hormone(TSH) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Measured in μU/mL
Change in free triiodothyronine (FT-3) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Measured in pg/mL
Change in free triiodothyronine (FT-3) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Measured in pg/mL
Change in free thyroxine (FT-4) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Measured in ng/mL
Change in free thyroxine (FT-4) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Measured in ng/mL
Change in white blood cell (WBC) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Measured in μ/L
Change in white blood cell (WBC) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Measured in μ/L
Change in platelet (PLT) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Measured in 10^4/μL
Change in platelet (PLT) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Measured in 10^4/μL
Change in bone age (BA) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Measured in year
Change in bone age (BA) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Measured in year
Change in bone age/chronological age (BA/CA) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Presented as ratio
Change in bone age/chronological age (BA/CA) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Presented as ratio
Change in electrocardiogram (ECG) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Assessment of change in ECG is measured by categories recorded in case report forms (CRFs): normal, abnormal not clinically significant and abnormal clinically significant.
Change in electrocardiogram (ECG) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Assessment of change in ECG is measured by categories recorded in CRFs: normal, abnormal not clinically significant and abnormal clinically significant.
Change in height standard deviation score (HSDS) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Presented as SD score
Change in height standard deviation score (HSDS) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Presented as SD score
Height velocity standard deviation score (HVSDS) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Presented as SD score
Height velocity standard deviation score (HVSDS) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Presented as SD score
Height velocity (HV) for non-naïve patients | Weeks 0, 52, 104, 156, 208, 260, 312, 364, 416, and 442 weeks
  Measured in cm/year
Height velocity (HV) for naïve patients | Weeks 0, 52, 104, 156, and 208 weeks
  Measured in cm/year

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (16):
- Japan (16):
  - Novo Nordisk Investigational Site, Asahikawa, Hokkaido
  - Novo Nordisk Investigational Site, Fukuoka
  - Novo Nordisk Investigational Site, Kanagawa
  - Novo Nordisk Investigational Site, Kyoto
  - Novo Nordisk Investigational Site, Maebashi-shi, Gunma
  - Novo Nordisk Investigational Site, Miyazaki
  - Novo Nordisk Investigational Site, Nagoya, Aichi
  - Novo Nordisk Investigational Site, Niigata-shi, Niigata
  - Novo Nordisk Investigational Site, Osaka
  - Novo Nordisk Investigational Site, Ōita
  - Novo Nordisk Investigational Site, Saitama-shi, Saitama
  - Novo Nordisk Investigational Site, Sapporo, Hokkaido
  - Novo Nordisk Investigational Site, Sendai-shi, Miyagi
  - Novo Nordisk Investigational Site, Shizuoka
  - Novo Nordisk Investigational Site, Tochigi
  - Novo Nordisk Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Muroya K, Kawai M, Yamagishi H, Endo T, Pietropoli A, Ferran JM, Horikawa R. Long-term effectiveness and safety of daily growth hormone therapy in Japanese children with Noonan syndrome: a post-marketing surveillance study. Endocr J. 2025 Nov 22. doi: 10.1507/endocrj.EJ25-0116. Online ahead of print. PMID 41285480